CLINICAL TRIAL: NCT05725213
Title: Non-interventional Study Investigating Photodynamic Therapy With Artificial Daylight Under Routine Clinical Conditions in Patients With Actinic Keratosis (ArtLight)
Brief Title: ADL-PDT Under Routine Clinical Conditions in Patients With Actinic Keratosis
Status: Completed | Type: Observational
Sponsor: Galderma Laboratorium GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: ArtLight
Record Dates: First submitted 2023-01-19; First posted 2023-02-13 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — methyl 5-aminolevulinate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Metvix® 160 mg/g Creme — Patients are treated with Metvix creme and exposed to artificial daylight
  Other Names: Methyl-5-aminolevulinate

SUMMARY:
The objective of this non-interventional study (NIS) is to gain comprehensive insights into the practicability of ADL-PDT with Metvix® in patients with actinic keratoses under real-world conditions.

DETAILED DESCRIPTION:
The objective of this non-interventional study (NIS) is to gain comprehensive insights into the practicability of ADL-PDT with Metvix® in patients with actinic keratoses under real-world conditions. Furthermore, this NIS will document the efficacy, satisfaction, safety and tolerability of ADL-PDT with Metvix® in routine use according to the label.

The observational study is designed as a multicenter study, covering all parts of Germany. Participating investigators are dermatologists experienced in ADL-PDT with an adequate pool of patients with actinic keratoses. The observation time per patient will comprise up to 6 months, including up to 4 visits.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study
* Age ≥18 years
* Thin or non-hyperkeratotic and non-pigmented actinic keratoses (AK) on the face or scalp (Olsen grade 1 or Olsen grade 2)
* The decision to undergo ADL-PDT with Metvix® was made independently of this study
* No contraindication (according to the SmPC)

Exclusion Criteria:

* Hypersensitivity to the active substance or to one of the other ingredients listed in section 6.1 of the SmPC or other ingredients, including peanut oil, peanut or soy.
* Morpheaform basal cell carcinoma
* Porphyria
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients selected from pool of dermatologists experienced in ADL-PDT with an adequate pool of patients with actinic keratoses.
Sampling Method: Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Real-world applicability of the ADL-PDT | 3 months after treatment
  Rate of resolved AK lesions in the focal region

SECONDARY OUTCOMES:
Change in skin quality over the course of the study overall and in the focus region | 3 months after treatment
  Change in skin quality over the course of the study overall and in the focus region through 5 scales questionnaire.
  Scale from 0 (none) to 5 (strong)
Change in AKASI score over the course of the study | 3 months after treatment
  Change in AKASI score over the course of the study Scale: 0 (no AK) to 18 (AK with highest level of severity)
Change in the number of lesions over the course of the study | 3 months after treatment
  Change in the number of lesions over the course of the study
Query of the type of skin preparation by the investigator | 3 months after treatment
  Query of the type skin preparation by the investigator through questionnaire.
Performance of artificial daylight exposure (artificial daylight system used) | 3 months after treatment
  Investigation which artificial daylight system is used through questionnaire.
Pain during and 5 min after artificial daylight exposure on a visual pain scale of 4 (moderate) to 10 (severe) | 3 months after treatment
  Pain during and 5 min after artificial daylight exposure on a visual pain scale of 4 (moderate) to 10 (severe)
Occurrence of local skin irritations or adverse events | 3 months after treatment
  Occurrence of local skin irritations or adverse events
Overall assessment of efficacy, tolerability, adherence, cosmetics by the investigator | 3 months after treatment
  Overall assessment (by investigator) of efficacy, tolerability, adherence, cosmetics through 5 scales questionnaire.
  Scale: 1 (very good) to 5 (very unsatisfied, or no effect at all)
Assessment of satisfaction by the patient | 3 months after treatment
  Assessment of satisfaction by the patient through questionnaire Scale: Very satisfied to very dissatisfied

CONTACTS AND LOCATIONS:
Overall Officials: Rolf-Markus Szeimies, Prof. Dr., Principal Investigator — KLINIKUM VEST GMBH - Knappschaftskrankenhaus Recklinghausen
Locations (1):
- Klinikum Vest GmbH, Recklinghausen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karrer S, Szeimies RM, Philipp-Dormston WG, Gerber PA, Prager W, Datz E, Zeman F, Muller K, Koller M. Repetitive Daylight Photodynamic Therapy versus Cryosurgery for Prevention of Actinic Keratoses in Photodamaged Facial Skin: A Prospective, Randomized Controlled Multicentre Two-armed Study. Acta Derm Venereol. 2021 Jan 4;101(1):adv00355. doi: 10.2340/00015555-3717. PMID 33313936